CLINICAL TRIAL: NCT05578677
Title: Endoscopic Biopsy Techniques in Barrett's Esophagus Patients
Acronym: BITE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Ilse Beaufort, Drs., St. Antonius Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: W21.022
Record Dates: First submitted 2022-01-07; First posted 2022-10-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Other): Single-biopsy advance-and-close
  Interventions: Other: Biopsy technique
- B (Other): Single-biopsy turn-and-suction
  Interventions: Other: Biopsy technique
- C (Other): Double-biopsy advance-and-close
  Interventions: Other: Biopsy technique
- D (Other): Double-biopsy turn-and-suction
  Interventions: Other: Biopsy technique

INTERVENTIONS:
Other: Biopsy technique — * Using the turn-and-suction technique, the forceps cups are opened and the forceps is withdrawn against the tip of the endoscope. The tip is then directed toward the target ('turn'), and suction is applied ('suction') as the forceps is applied against the targeted mucosa and then closed.
  * Endoscopists can obtain two biopsy specimens from a single passage of the conventional biopsy forceps instead of one. These techniques are called the 'double-biopsy method' and the 'single-biopsy method', respectively.

SUMMARY:
Barrett's esophagus (BE) is a premalignant condition of the distal esophagus, predisposing to dysplasia and esophageal adenocarcinoma. Therefore, in BE patients, current guidelines recommend endoscopic surveillance with four-quadrant biopsies every 2 centimeters of the Barrett's length. These biopsies need to be of optimal quality for adequate histopathological assessment. Larger biopsies can facilitate adequate histopathological assessment because (1) more tissue is available, (2) larger biopsies usually result in less superficial biopsies, with all mucosal layers present in the biopsy specimen, and (3) larger biopsies will ease orientation of the specimen. In a pilot study, the investigators found a median increase of nearly 30% in surface area when the biopsies were obtained by BE-expert endoscopists in comparison with non BE-expert endoscopists. A possible explanation for this difference can be biopsy method or technique. BE-expert endoscopists use the single biopsy method and turn-and-suction technique, whereas the double biopsy method and the advance-and-close technique are the more generally used biopsy techniques within non BE-expert endoscopists.

The BITE study is therefore designed to identify the preferred biopsy technique and method in BE patients in order to optimise biopsy quality and histopathological assessment.

DETAILED DESCRIPTION:
This study will consist of three consecutive parts: a retrospective analysis, a two-by-two factorial randomised study, and a prospective before after study. The results of the preceding part of the BITE study will determine the continuation with subsequent part. If the second part of the BITE-study fails to identify a specific technique as the optimal biopsy technique (i.e. biopsy size is not significantly increased by using the single-biopsy turn-and-suction technique), the investigators will not proceed with the third step of the BITE-study.

Part I - retrospective analysis The retrospective analysis will be performed. This analysis of biopsy size aims to properly compare biopsy size of esophageal biopsies taken by BE-expert en non-expert endoscopists.

Part II - Two-by-two factorial design randomised study The second part of the BITE study is a two-by-two factorial design randomised study. This is a prospective, individually randomised study and will be performed in two different hospitals in the Netherlands: St. Antonius Hospital Nieuwegein and University Medical Centre Utrecht (UMCU). Patients who are willing to participate will be randomised into four different groups: in group A, biopsies will be taken using the single-biopsy advance-and-close technique; in group B, biopsies are obtained by the single-biopsy turn-and-suction technique; in group C the double-biopsy advance-and-close technique will be used; and group D, biopsies will be taken by the double-biopsy turn-and-suction technique. All upper endoscopies will be performed by BE-expert endoscopists.

Part III - retrospective before-after study The third and last part of the BITE study is a prospective before-after study. If the single-biopsy turn-and-suction technique proves to be the superior biopsy technique, this technique will be implemented among non BE-expert endoscopists. Non BE-expert endoscopists will be trained in the turn-and-suction technique, and data will be collected of biopsies before and after the training. If the second part of the BITE-study fails to identify the single-biopsy turn-and-suction technique as the optimal biopsy technique (i.e. biopsy size is not significantly increased by using the single-biopsy turn-and-suction technique), the investigators will not proceed with the third step of the BITE-study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* A diagnosis of Barrett's esophagus (maximum length ≥ 1cm)
* Scheduled for surveillance endoscopy with random biopsies
* In addition to the abovementioned inclusion criteria, a subject must meet the following criteria to participate in:

Part I: endoscopy performed by BE expert or non-BE expert endoscopists Part II: endoscopy performed by BE expert endoscopist Part III: endoscopy performed by non-BE expert endoscopist

Exclusion Criteria:

* Very long BE segment (maximum length ≥ 10cm)
* Any known clinical contraindication for obtaining biopsies (e.g. oesophageal varices, uncontrolled coagulopathy)
* Biopsies of suspicious lesions in the Barrett's epithelium will be excluded from analysis in all parts of this study. In case of suspicious lesions, endoscopists (in part II and part III of the BITE study) are allowed to obtain biopsies according to the technique they prefer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Size of biopsy specimen, as assessed by a blinded study investigator | 14 days
  Surface area of biopsy specimen in mm2

SECONDARY OUTCOMES:
The percentage of biopsies in which the muscularis mucosae is present as assessed by a blinded upper GI-pathologist | 14 days
  Muscularis mucosa present, only strands of muscularis mucosa present, muscularis mucosa absent.
The percentage of biopsies with the presence of crush artefacts in the biopsy specimen, as assessed by a blinded upper GI-pathologist | 14 days
  Absent, <50% of the biopsy specimen, or >50% of the biopsy specimen
The number of lost biopsy specimens, as assessed by the endoscopy nurse | Day 0, during the endoscopy
  The number of times two biopsies have been taken, and only one biopsy specimen is present in the container that is sent to the pathology department
The total biopsy time, as assessed by the endoscopy nurse | Day 0, during the endoscopy
  Time between first insertion of the biopsy forceps until the last biopsy specimen has reached the jar, divided by the number of biopsies per patient
The percentage biopsies with the presence of dysplasia, as assessed by a blinded upper GI pathologist | 14 days
  The presence of dysplasia in biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: B. Weusten, prof. Dr., Principal Investigator — St. Antonius Hospital; B. Weusten, prof. Dr., Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No